CLINICAL TRIAL: NCT05166369
Title: Optimisation of Antibiotic Prescription in Acute Non-complicated Respiratory Tract Infections in Children: a Multicenter Factorial Randomised Controlled Trial Targeting Health Professionals and Parents.
Brief Title: Optimisation of Antibiotic Prescription in Acute Noncomplicated Respiratory Tract Infections in Children (OptimAP Study)
Acronym: OptimAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Fundació La Marató de TV3 (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 19/019-P
Record Dates: First submitted 2021-11-24; First posted 2021-12-21 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Acute Respiratory Tract Infections
Keywords: Acute respiratory tract infection; Microbial Antibiotic Resistance; Communication skills training; Mobile app-based health information and education

STUDY DESIGN:
Intervention Model Description: Multicenter, cluster, randomized, factorial, controlled trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Intervention targeted to healthcare providers (paediatricians, nurses and pharmacists) (ITHP) (Experimental): Professionals in the PC centres allocated to this group will receive a complex intervention, delivered remotely, which will include the following components:
  i) Web based training that will include: communication skills training and optimal management of acute non-complicated RTI, including a specific training on delayed antibiotic prescription.
  ii) By-monthly feedback about the rate of antibiotic prescription and consumption for RTI, center level and individual pediatrician level (information automatically gathered from electronic health records).
  Interventions: Behavioral: Communication skills training
- Intervention targeted to parents (ITP) (Experimental): PC centres allocated to this group will display posters and flyers to inform parents and/or caregivers about a mobile app. It will provide detailed information about respiratory tract infections and optimal use of antibiotics. The app will include information that will be of use before the consultation, but it will also allow the patient to interact with the physician during the consultation, potentially improving share decision-making. Importantly, the app will allow tailoring the guidance provided according to the type of infection or number of days with symptoms. The app will be accessible through an app store or directly using a QR (quick response) code to facilitate uptake. Professionals in the primary care centres allocated to this group will also receive a by-monthly feedback about the rate of antibiotic prescription and consumption for RTI, at center level and individual pediatrician level (information automatically gathered from electronic health records).
  Interventions: Behavioral: Mobile phone application on RTI
- Intervention targeted to patients and/or patient´s parents and to the healthcare providers (ITHP*P) (Experimental): Centres allocated to this group will receive the two interventions described above (intervention targeted to parents plus intervention targeted to providers).
  Interventions: Behavioral: Communication skills training; Behavioral: Mobile phone application on RTI
- Control group (No Intervention): The centers allocated to this arm of the study will continue with their usual care. To avoid a potential Hawthorne effect (observer effect) these centers will not be informed about their participation as controls.

INTERVENTIONS:
Behavioral: Communication skills training — This intervention consists of a course on communication skills for healthcare professionals.
  It will be done remotely via the internet and will include: communication skills training and optimal management of acute non-complicated RTI and delayed antibiotic prescription. Training modules will be delivered via a specific website password protected. Healthcare professionals will also receive a by-monthly feedback about the rate of antibiotic prescription and consumption for RTI.
  Arms: Intervention targeted to healthcare providers (paediatricians, nurses and pharmacists) (ITHP); Intervention targeted to patients and/or patient´s parents and to the healthcare providers (ITHP*P)
Behavioral: Mobile phone application on RTI — This intervention involves the use of a mobile phone application by parents and caregivers.
  The mobile app will provide information, education and interactive tools about acute noncomplicated respiratory tract infections.
  PC centres allocated to this group will display posters and flyers to inform parents and caregivers about the mobile app. Healthcare staff will also promote the use of this app by parents and caregivers.
  The app information will be useful before the consultation, and will also allow the patient to interact with the physician during the consultation, potentially improving share decision-making.
  Importantly, the app will allow tailoring the guidance provided according to the type of infection or the number of days with symptoms.
  Healthcare professionals in the primary care centres allocated to this group will also receive a by-monthly feedback about the rate of antibiotic prescription and consumption for RTI.
  Arms: Intervention targeted to parents (ITP); Intervention targeted to patients and/or patient´s parents and to the healthcare providers (ITHP*P)

SUMMARY:
Background: High-volume antibiotic prescribing in primary care is a major driver of antibiotic resistance. Education of physicians and patients can lower prescribing levels, but it frequently relies on highly trained staff. We will assess whether remotely delivered complex interventions including internet-based training for health care provider, and an educational intervention for parents could improve prescribing practices for respiratory tract infections (RTI) in Spain.

Methods: We will develop and evaluate the feasibility of two interventions in a 16-months randomized controlled factorial trial. Primary care (PC) centres will be allocated to one of the following four groups:

1. Intervention targeting healthcare providers (paediatricians, nurses and pharmacists): i) Internet based training about communication skills and optimal antibiotic prescribing (including delayed prescribing); ii) bimonthly antibiotic prescription feedback.
2. Intervention targeting parents: PC centres allocated to this group will display posters and flyers presenting a mobile app that will include information about respiratory tract infections and optimal use of antibiotics. The app can be used before, during and after the consultation, providing condition specific and patient tailored information.
3. Intervention targeting both providers and parents
4. No intervention.

During the trial duration we will conduct a process evaluation and a cost-effectiveness analysis. Our primary outcome will be change in the total antibiotic prescription rate. Our secondary outcomes will include: respiratory complications (e.g. pneumonia), antibiotic related adverse effects, repeated consultations, and antibiotic consumption in relation with antibiotic prescribing (delayed antibiotic prescribing). Assuming an average cluster size of 200 RTI consultations per centre, we will need to recruit 222 PC centres.

DETAILED DESCRIPTION:
This project will evaluate the effectiveness of two complex interventions to optimize the use of antibiotics in acute uncomplicated respiratory tract infections (RTI). We will first develop the different components of the interventions and evaluate their feasibility (user testing). We will then conduct a multicenter, randomized, controlled trial to evaluate the effectiveness of the overall intervention and its two main constituents in reducing antibiotic consumption. For this reason we will implement a 2x2 factorial randomized cluster clinical trial based on healthcare practices. They will be randomized to receive the intervention targeted to parents, intervention targeted health care professionals, both interventions, or none of them. We will need to recruit a sample size of 222 primary care centres, allocated in a ratio of 1:1:1:1 to one of the four intervention groups (assuming an average cluster size of 200 RTI consultations per centre). Study setting will be defined as primary care centres in four Autonomous Communities in Spain (Catalonia, Balearic Islands, Navarra and Basque Country) with a total of more than 600 PC centers, 1,200 pediatricians, and more of one million children. Finally, during the trial duration, we will conduct a process evaluation and an economic evaluation with a cost-effectiveness analysis.

The interventions include the main characteristics of successful interventions to reduce antibiotic prescribing identified in a systematic review: engage children, occur prior to an illness episode, employ delayed prescribing, and provide guidance on specific symptoms (Andrews 2012). Furthermore, the factorial design will inform about their relative merits and the process evaluation about the potential effect of the individual components.

The research team in in Barcelona (Spain) will coordinate the overall running of the project. A research coordinator in Barcelona will run the day to day of the project from day one under the supervision of the principal investigator. The research teams in four different Spanish Autonomous Communities will contribute to all the stages (intervention development, clinical trial, and economic and process evaluation). Patient representatives will be involved in the project as co-investigators and members of the Steering Committee. Throughout the project groups of parents at each of the regions will be providing feedback.

ELIGIBILITY:
Inclusion Criteria:

* Healthcare professionals who care for children in primary care centres and community pharmacists of reference in four Autonomous Communities of Spain (Catalonia, Balearic Islands, Navarra and Basque Country).

Exclusion Criteria:

* None

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 222 (Actual)
Dates: Start 2022-01-03 (Actual); Primary Completion 2023-09-04 (Actual); Study Completion 2023-09-05 (Actual)

PRIMARY OUTCOMES:
Total antibiotic prescription rate | Three months (from 1st January 2022 to 31st March 2022)
  Total antibiotic prescription rate for patients between 0 and 14 years old (children).

SECONDARY OUTCOMES:
RTI complication rate | Three months (from 1st January 2022 to 31st March 2022)
  Rate of clinical complications of respiratory tract infection (e.g. pneumonia, otitis media, sinusitis).
Hospital admission rate due to RTI | Three months (from 1st January 2022 to 31st March 2022)
  Hospital admission rate due to a RTI or a related complication at 30 days after index RTI consultation.
RTI Re-consultation rate | Three months (from 1st January 2022 to 31st March 2022)
  RTI re-consultations rates at 7, 14, or 31 days after index RTI consultation.
Antibiotic-related adverse events rate | Three months (from 1st January 2022 to 31st March 2022)
  Antibiotic-related adverse events rate (as registered in clinical records).

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Alonso Coello, PhD, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau
Locations (4):
- Spain (4):
  - Institut d'Investigació de les Illes Balears (IdISBa), Palma de Mallorca, Balearic Islands
  - Osakidetza - Ambulatorio de Pasai San Pedro, Pasaia, Gipuzkoa
  - Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau, Barcelona
  - Servicio Navarro de Salud - Osasunbidea, Pamplona

IPD SHARING:
Plan to Share IPD: Yes
There is not specific individual participant data, but primary care centre data sets.
Supporting Information: Study Protocol, SAP, ICF, CSR

REFERENCES:
- [Result] Andrews T, Thompson M, Buckley DI, Heneghan C, Deyo R, Redmond N, Lucas PJ, Blair PS, Hay AD. Interventions to influence consulting and antibiotic use for acute respiratory tract infections in children: a systematic review and meta-analysis. PLoS One. 2012;7(1):e30334. doi: 10.1371/journal.pone.0030334. Epub 2012 Jan 27. PMID 22299036
- [Result] Costelloe C, Metcalfe C, Lovering A, Mant D, Hay AD. Effect of antibiotic prescribing in primary care on antimicrobial resistance in individual patients: systematic review and meta-analysis. BMJ. 2010 May 18;340:c2096. doi: 10.1136/bmj.c2096. PMID 20483949
- [Result] Ranji SR, Steinman MA, Shojania KG, Gonzales R. Interventions to reduce unnecessary antibiotic prescribing: a systematic review and quantitative analysis. Med Care. 2008 Aug;46(8):847-62. doi: 10.1097/MLR.0b013e318178eabd. PMID 18665065
- [Result] Little P, Stuart B, Francis N, Douglas E, Tonkin-Crine S, Anthierens S, Cals JW, Melbye H, Santer M, Moore M, Coenen S, Butler C, Hood K, Kelly M, Godycki-Cwirko M, Mierzecki A, Torres A, Llor C, Davies M, Mullee M, O'Reilly G, van der Velden A, Geraghty AW, Goossens H, Verheij T, Yardley L; GRACE consortium. Effects of internet-based training on antibiotic prescribing rates for acute respiratory-tract infections: a multinational, cluster, randomised, factorial, controlled trial. Lancet. 2013 Oct 5;382(9899):1175-82. doi: 10.1016/S0140-6736(13)60994-0. Epub 2013 Jul 31. PMID 23915885